CLINICAL TRIAL: NCT01022359
Title: Comparison of Tesio and LifeCath Twin Permanent Dialysis Catheters
Acronym: VyTes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08/H0710/24
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: Hemodialysis
Keywords: haemodialysis; vascular access; central venous catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tesio Catheter (Active Comparator): Patients randomised to receive the established catheter type in use at our centre [control]
  Interventions: Device: TesioCath
- LifeCath (Active Comparator): Patients randomised to receive the LifeCath Twin catheter - the catheter type being compared to the standard line in use at our centre (Tesio)
  Interventions: Device: LifeCath Twin

INTERVENTIONS:
Device: TesioCath — Insertion of the TesioCath(TM) central venous catheter for haemodialysis vascular access
  Other Names: BioFlex TesioCath (TM) - MedComp, Harleysville, PA, USA
  Arms: Tesio Catheter
Device: LifeCath Twin — Insertion of the LifeCath Twin central venous catheter for haemodialysis vascular access
  Other Names: Vygon LifeCath Twin - Vygon(UK) Ltd, Cirencester, Gloucs, UK
  Arms: LifeCath

SUMMARY:
This study aims to compare two available types of central venous haemodialysis catheters (lines) - CVCs, and will examine how easy they are to insert, complications, blood flow on dialysis over time, line loss, line clotting and infective events. It will examine whether the LifeCath type of CVC can deliver high blood flow rates from first use after insertion and equivalent function and complication rate to the Tesio type of CVC that is in use in our centre already. Complications relating to dialysis access make up 30% of admissions for haemodialysis patients and so this is a study that could benefit patients and their care providers.

DETAILED DESCRIPTION:
Complications relating to dialysis access make up to 30% of admissions in haemodialysis patients. Comparative studies of complications between dialysis lines can help physicians and patients choose the best CVC type. In addition determining a type of dialysis line that can deliver good blood flows from the outset can minimise length of hospital stay for access creation. This study aims to perform a head-to-head comparison of two very similar (twin catheter) dialysis lines and examine short and long-term function as well as complication rates at our centre.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* No history of prior central venous catheter insertion
* Medically fit for procedure (able to lie flat, no haemodynamic instability)
* No active infection (recent positive blood cultures, clinical signs of infection, CRP>100)
* Able to give informed consent
* Expected to survive more than 12 months after catheter insertion

Exclusion Criteria:

* As above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neill Duncan, MBBS MRCP, Principal Investigator — Imperial College Healthcare NHS Trust; Albert Power, MBBChir MRCP, Study Director — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Duncan ND, Singh S, Cairns TD, Clark M, El-Tayar A, Griffith M, Hakim N, Hamady M, McLean AG, Papalois V, Palmer A, Taube D. Tesio-Caths provide effective and safe long-term vascular access. Nephrol Dial Transplant. 2004 Nov;19(11):2816-22. doi: 10.1093/ndt/gfh467. Epub 2004 Aug 31. PMID 15340094
- [Background] Perini S, LaBerge JM, Pearl JM, Santiestiban HL, Ives HE, Omachi RS, Graber M, Wilson MW, Marder SR, Don BR, Kerlan RK Jr, Gordon RL. Tesio catheter: radiologically guided placement, mechanical performance, and adequacy of delivered dialysis. Radiology. 2000 Apr;215(1):129-37. doi: 10.1148/radiology.215.1.r00mr43129. PMID 10751478
- [Background] Hassell DD 3rd, Vesely TM, Pilgram TK, Audrain JL. Initial performance of Tesio hemodialysis catheters. J Vasc Interv Radiol. 1999 May;10(5):553-8. doi: 10.1016/s1051-0443(99)70082-5. PMID 10357479
- [Result] Power A, Hill P, Singh SK, Ashby D, Taube D, Duncan N. Comparison of Tesio and LifeCath twin permanent hemodialysis catheters: the VyTes randomized trial. J Vasc Access. 2014 Mar-Apr;15(2):108-15. doi: 10.5301/jva.5000202. Epub 2014 Feb 5. PMID 24500851

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tesio Catheter | LifeCath
Started | 39 | 41
Completed | 39 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tesio Catheter | LifeCath | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (15.6) | 58.9 (16.4) | 61 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 29 | 26 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Blood Flow Rate at First Use After Insertion
Time Frame: First haemodialysis session after insertion
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Tesio Catheter | LifeCath
Number analyzed (Participants) | 39 | 41
mL/min | 277 (79) | 383 (82)

2. Secondary Outcome: Achievement of Flow Rates>=450ml/Min at Dialysis Session
Time Frame: flow rate measured at each session; session at 12 months reported
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Tesio Catheter | LifeCath
Number analyzed (Participants) | 39 | 41
mL/min | 361 (48) | 379 (43)

3. Secondary Outcome: Line Retention (Either/Both Lumens)
Time Frame: 12 months
Population: measure not taken
Arm/Group | Tesio Catheter | LifeCath
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Infective Episodes (Catheter & Non-catheter Related)
Time Frame: 12 months
Population: measure not collected
Arm/Group | Tesio Catheter | LifeCath
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Catheter Dysfunction Requiring Use of Thrombolytic Agents
Time Frame: 12 months
Measure: Number; unit: thrombolytic infusions
Arm/Group | Tesio Catheter | LifeCath
Number analyzed (Participants) | 39 | 41
thrombolytic infusions | 0 | 6

6. Secondary Outcome: Complications at Catheter Insertion
Time Frame: Day 1
Measure: Number; unit: complications at insertion
Arm/Group | Tesio Catheter | LifeCath
Number analyzed (Participants) | 39 | 41
complications at insertion | 0 | 0

7. Secondary Outcome: Recirculation Rates
Time Frame: 12 months
Population: measure not taken
Arm/Group | Tesio Catheter | LifeCath
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of trial, 12 months
Arm/Group | Tesio Catheter | LifeCath
All-Cause Mortality (participants affected / at risk) | 3/39 | 4/41
Serious Adverse Events (participants affected / at risk) | 3/39 | 4/41
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tesio Catheter (N=39) | LifeCath (N=41)
sudden cardiac death (Cardiac disorders) | 0 (0) | 2 (2)
myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
pulmonary sepsis (Cardiac disorders) | 0 (0) | 1 (1)
severe hemorrhagic stroke (Cardiac disorders) | 1 (1) | 0 (0)
metastatic malignancy that was diagnosed 9 months following CVC insertion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes